CLINICAL TRIAL: NCT00278109
Title: Phase I/II Partial Breast Irradiation With Concurrent Chemotherapy
Brief Title: Partial Breast Irradiation With Chemotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0381; P30CA006973 (NIH); CDR0000446085; 04-03-22-01 (Other: JHM IRB)
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Results first posted 2019-03-28 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Doxorubicin; Radiation

ARMS (1):
- PBI with Concurrent Chemotherapy (Experimental): Phase I Single Arm study of PBI with concurrent chemotherapy. Primary endpoint is radiation toxicity. The intervention is partial breast radiation with doxorubicin and cyclophosphamide.
  Interventions: Drug: cyclophosphamide; Drug: Doxorubicin; Radiation: radiation

INTERVENTIONS:
Drug: cyclophosphamide — chemotherapy
  Other Names: adriamycin
Drug: Doxorubicin — doxorubicin
  Other Names: cytoxan
Radiation: radiation — radiation

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as cyclophosphamide and doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy together with cyclophosphamide and doxorubicin after surgery may kill any tumor cells that remain.

PURPOSE: This phase I/II trial is studying the side effects of radiation therapy when given together with cyclophosphamide and doxorubicin and to see how well they work in treating women with stage I or stage II breast cancer who have undergone surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the potential acute and late skin and subcutaneous toxicities in women with resected stage I or II breast cancer treated with partial breast irradiation (PBI) and concurrent cyclophosphamide/doxorubicin (AC) chemotherapy.
* Assess the cosmetic effects of partial breast irradiation/chemotherapy (PBIC) in these patients.
* Assess the local control rate in patients treated with this regimen.

OUTLINE: Patients undergo partial breast radiotherapy once daily, 5 days a week, for 3 weeks. Patients also receive doxorubicin IV over 15 minutes and cyclophosphamide IV over 30 minutes on day 1. Treatment with doxorubicin and cyclophosphamide repeats every 2 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for approximately 10 years.

PROJECTED ACCRUAL: A total of 42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast by routine hematoxylin and eosin (H&E) staining

  * Primary tumor ≤ 4 cm and 0-3 positive axillary lymph nodes (pathologic T1-2, pathologic N0-N1, M0)

    * Patients with lymph nodes positive only by cytokeratin staining (i.e., H&E negative) are eligible
* No squamous cell carcinoma or sarcoma of the breast
* Patients must have undergone a segmental mastectomy (SM) with a level I and ll axillary dissection or sentinel lymph node biopsy within the past 14 weeks

  * Surgical margins at the time of SM must be negative (> 3 mm) for both invasive carcinoma and for non-invasive ductal carcinoma
* No active local-regional disease
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Sex: female
* Menopausal status not specified
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective non-hormonal contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No other serious or poorly controlled medical or psychiatric condition that could be exacerbated by, or complicate compliance with study treatment

PRIOR CONCURRENT THERAPY:

* No prior radiation therapy to the breast
* No prior trastuzumab (Herceptin ®)
* No other concurrent chemotherapy
* No concurrent hormonal therapy except the following:

  * Steroids given for adrenal failure
  * Hormones administered for non-disease-related conditions (e.g., insulin for diabetes, synthroid for hypothyroidism)
  * Intermittent dexamethasone as an antiemetic or premedication

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2004-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard C. Zellars, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Jean Wright, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] Zellars RC, Frassica D, Stearns V, et al.: Phase I/II trial of partial breast irradiation with concurrent dose-dense doxorubicin and cyclophosphamide (ddAC) chemotherapy in early stage breast cancer: report of skin toxicity and cosmetic outcome. [Abstract] Int J Radiat Oncol Biol Phys 69 (3 Suppl): A-44, S26, 2007.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two patients did not initiate study procedures: one was found to have residual gross disease during treatment planning, and another withdrew consent.
Groups:
- Experimental: cyclophosphamide: chemotherapy
  doxorubicin hydrochloride: chemotherapy
  adjuvant therapy: chemotherapy
  radiation therapy: chemotherapy
Period: Overall Study
Arm/Group | Experimental
Started | 25
Completed 3 Cycles of Chemotherapy | 25
Completed | 21
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — social circumstances | 1

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 25
Age, Customized [Count of Participants; unit: Participants]
  Age <= 45 years | 5
  Age >= 45 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Acute, Late Skin, and Subcutaneous Toxicity
Description: Number of participants with Grade 4 toxicity as defined by the following criteria:
  Acute Skin Toxicity: 0=No change, 1= Follicular, faint, or dull erythema/epilation/dry/desquamation/decreased swelling, 2= Tender or bright erythemal patchy moist desquamation/moderate edema, 3= Confluent moist desquamation other than skin folds, piting edema, 4= Ulceration, hemorrahage, necrosis, Late Skin Toxicity: 0= None, 1= Slight Atrophy, Pigmentation change, some hair loss, 2= Patch atrophy, moderate telangectasias, total hair loss, 3= Marked atrophy, gross telangectasias, 4= Ulceration; Subcutaneous Tissue Toxicity: 0= None, 1= Slight induration (fibrosis) and loss of subcutaneous fat, 2= Moderate fibrosis but asymptomatic; slight field contracture; <10% linear reduction, 3= Severe induration and loss subcutaneous tissue; field contracture >10% linear reduction; 4= Necrosis
Time Frame: up to 5 years
Population: Data was only collected on participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 25
Participants | 0

ADVERSE EVENTS:
Time Frame: Weekly then monthly then annually for up to 5 years.
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 21/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=25)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=25)
perianal dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
foot blisters (Skin and subcutaneous tissue disorders) | 1 (1)
cough/bronchospasms (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Absolute neutrophil count (Blood and lymphatic system disorders) | 4 (4)
Nausea & vomiting (Gastrointestinal disorders) | 3 (3)
Mucositis (Immune system disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Contralateral breast abscess (Infections and infestations) | 1 (1)
Grade 1 Radiation Dermatitis (Skin and subcutaneous tissue disorders) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No